CLINICAL TRIAL: NCT03941795
Title: A Randomized, Controlled, Multicenter Phase II Clinical Study to Evaluate the Efficacy and Safety of Toripalimab Injection Combined With Axitinib in the First-Line Treatment of Patients With Advanced Mucosal Melanoma
Brief Title: Phase II Study in the Treatment of Patients With Advanced Mucinous Melanoma
Acronym: BJCH-MM-0624
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-MM-0624
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Advanced Mucosal Melanoma
Keywords: PD-1 monoclonal antibody; the First Line Therapy; Axitinib; Mucosal Melanoma; Toripalimab; JS001
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JS001(Toripalimab Injection) Combined With Axitinib (Experimental)
  Interventions: Other: JS001 and Axitinib
- JS001 alone (Experimental)
  Interventions: Biological: JS001(Toripalimab Injection)
- Axitinib alone (Active Comparator)
  Interventions: Drug: Axitinib 1 MG [Inlyta]

INTERVENTIONS:
Biological: JS001(Toripalimab Injection) — Test Group:
  Toripalimab (240 mg, IV, Q3W) + axitinib (5 mg/tablet, one tablet, twice a day, orally); axitinib is started on the second day of administration of toripalimab until disease progression or intolerable toxicity, the investigator or subject decides to withdraw, lost to follow-up, initiation of other antineoplastic therapy, or death, with a maximum duration of toripalimab use of no more than 2 years.
  Arms: JS001 alone
Drug: Axitinib 1 MG [Inlyta] — Axitinib (5 mg/tablet) one tablet, twice a day, orally until disease progression or intolerable toxicity, the investigator or subject decides to withdraw, lost to follow-up, initiation of other antineoplastic therapy, or death
  Arms: Axitinib alone
Other: JS001 and Axitinib — Control Group:
  Toripalimab (240 mg, IV, Q3W) is administered on the first day until disease progression or intolerable toxicity, the investigator or subject decides to withdraw, lost to follow-up, initiation of other antineoplastic therapy, or death, with a maximum duration of no more than 2 years
  Arms: JS001(Toripalimab Injection) Combined With Axitinib

SUMMARY:
This is a randomized, controlled, multicenter Phase II clinical study to evaluate the efficacy and safety of toripalimab injection combined with axitinib in the first-line treatment of patients with advanced mucosal melanoma. The target population is the patients with previously untreated, histopathologically confirmed, unresectable or metastatic mucosal melanoma. At the randomization, patients are randomized 1:1:1 into three groups with approximately 33 subjects in each group to receive toripalimab injection plus axitinib, toripalimab injection monotherapy (subjects who meet the criteria after disease progression may cross over to receive toripalimab plus axitinib), or axitinib monotherapy (subjects who meet the criteria after disease progression may cross over to receive toripalimab plus axitinib); when the patient has disease progression or intolerable toxicity, the treatment is terminated, and the survival follow-up will be initiated.

ELIGIBILITY:
Inclusion Criteria Patients are eligible for the trial if they meet the following criteria:

1. Men and women, aged 18 to 80 years.
2. Patients with pathohistologically confirmed, unresectable or metastatic mucosal melanoma.
3. No prior treatment with any systemic antineoplastic agents (prior adjuvant or neoadjuvant therapy is allowed, but should be completed at least 3 weeks prior to randomization and all related adverse events have returned to normal or CTC-AE Grade 1).
4. Have a score of 0 or 1 on the ECOG scale.
5. Tumor tissue samples must be available for PD-L1 expression testing.
6. At least one measurable lesion according to RECIST 1.1, and the lesion has not been irradiated.
7. Organ function must meet the following requirements (within 7 days prior to randomization):

   Peripheral blood: absolute neutrophil count (ANC) ≥1.5 × 109/L, platelets (PLT) ≥100 × 109/L, hemoglobin (HB) ≥9 g/dL (no blood transfusion or blood components within 14 days before testing); Liver: Serum bilirubin (TBIL) ≤1.5 x upper limit of normal (ULN),, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x ULN (≤5 x ULN in case of liver metastases); Serum creatinine ≤1.5 x ULN; International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5 x ULN (only for patients not receiving anticoagulant therapy; patients receiving anticoagulant therapy should keep the anticoagulant within the therapeutic requirements); Normal cardiac function, i.e., normal or abnormal electrocardiogram without clinical significance, and left ventricular ejection fraction (LVEF) greater than 50% on cardiac ultrasound.
8. Women of childbearing age must have a negative pregnancy test within 7 days prior to treatment; men of reproductive potential or women of childbearing potential must use highly effective contraceptive methods (e.g., oral contraceptives, intrauterine contraceptive devices, abstinence or barrier contraception in combination with spermicides) throughout the trial and continue contraception for 3 months after the end of treatment.
9. Subjects are willing to participate in this study and sign informed consent form, have good compliance and cooperate with the follow-up.

Exclusion Criteria Patients with any of the following conditions will be excluded from the trial:

1. Patients previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2 therapy and/or VEGFR TKIs.
2. Patients who have participated in or are participating in clinical trial of other drug/therapy within 4 weeks prior to this study treatment (before randomization).
3. Major surgery, live vaccination, immunotherapy within 4 weeks prior to study start, and radiotherapy within 2 weeks prior to study start.
4. History of malignancy other than mucosal melanoma within the past 3 years, with the exception of cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early stage prostate cancer, and carcinoma in situ of the cervix.
5. Patients who received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF) and erythropoietin, within 1 week prior to study start.
6. HIV test positive.
7. Patients with active hepatitis B or C:

   * If HBsAg or HBcAb is positive, additionally test HBV DNA (results above the lower limit of detection at site);
   * If the result of HCV antibody test is positive, additionally test HCV RNA.
8. Known to be allergic to recombinant humanized PD-1 monoclonal antibody drug and its components; known to be allergic to axitinib and any of its excipients.
9. Hypertension that cannot be controlled by medication.
10. Massive pleural effusion or ascites with clinical symptoms requiring symptomatic management.
11. Subjects with active central nervous system (CNS) metastases are excluded. Subjects with metastatic brain lesions are eligible if they have received treatment and have no evidence of disease progression on magnetic resonance imaging (MRI) at least 8 weeks after completion of treatment and within 28 days before the first dose. Immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalent) must not be required at least 2 weeks prior to study drug administration.
12. History of active pulmonary tuberculosis.
13. Have any uncontrollable clinical problems, including but not limited to:

    * Active autoimmune disease requiring systemic steroid/immunosuppressive therapy, such as hypophysitis, colitis, hepatitis, nephritis, etc.;
    * Have the following occurrence within 6 months prior to randomization: 1) deep vein thrombosis or pulmonary embolism; 2) percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; 3) cerebrovascular accident, transient ischemic attack.
    * Other serious, uncontrollable concomitant illness that may affect protocol compliance or interfere with interpretation of results, including active opportunistic infection or progressive (severe) infection, uncontrolled diabetes, cardiovascular disease (New York Heart Association class III or IV heart failure, second degree or higher heart block, myocardial infarction within the past 6 months, unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc.) or pulmonary disease (history of interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm).
14. Any condition that affects the subject's swallowing of the drug, and any condition that affects the absorption or pharmacokinetics of the investigational product.
15. Have received stem cell transplant or organ transplant.
16. Women of childbearing age, pregnant or lactating women with positive serum or urine pregnancy test 7 days before starting treatment.
17. Have a history of psychotropic drug abuse and unable to withdraw or have a history of mental disorders.
18. Other severe, acute, or chronic medical conditions or laboratory abnormalities that, in the judgment of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
19. Patients who are judged by the investigator to have poor compliance, or other conditions that make them unsuitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the progression-free survival (PFS) | 36 months
  Progression-free survival (PFS) per RECIST 1.1 criteria: Time from the date of randomization to the first documented disease progression (per RECIST 1.1 criteria), or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
INV-ORR | 36 months
  INV-ORR in crossover subjects is the number of subjects with DOR of CR or PR based on INV assessment divided by the number of crossover subjects. DOR is defined as the best response recorded as measured by INV from the date of the first crossover dose to the date of objective documentation of progression per RECIST 1.1 or the date of subsequent therapy, including tumor-directed radiotherapy and tumor-directed surgery, whichever occurs first. For subjects without documented progression or subsequent treatment, all available response designations will be assigned to the DOR evaluation. Baseline tumor assessments for crossover subjects are based on the last tumor assessment for monotherapy prior to the combination crossover. Exploratory endpoints will be analyzed at the time of primary endpoint analysis if data are available.
ORR | 36 months
  Objective response rate (ORR) according to RECIST 1.1;
PFS | 36 months
  Progression-free survival (PFS) according to RECIST 1.1;
DOR | 36 months
  Duration of response (DOR) according to RECIST 1.1;
TTR | 36 months
  Time to response (TTR) according to RECIST 1.1;
DCR | 36 months
  Disease control rate (DCR) according to RECIST 1.1;
OS | 36 months
  Overall survival (OS): Time from the date of randomization to death from any cause. Surviving patients as of the date of analysis will be censored at the date of their last contact.
safety: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 36 months
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD,PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Baishen First Hospital of Jilin University, Shengyang, Liaoning